CLINICAL TRIAL: NCT00404040
Title: A Single Centre Study to Assess the Safety and Efficacy of Movicol in the Treatment of Faecal Impaction in Children Followed by a Double Blind, Randomised Phase to Compare the Safety and Efficacy of Movicol and Lactulose for Maintenance Therapy
Brief Title: Movicol in Childhood Constipation (ProMotion Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 99/05 (Part II)
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — Lactulose

INTERVENTIONS:
Drug: Polyethylene glycol 3350 NA bicarbonate NaCl KCl (Movicol)
Drug: Lactulose

SUMMARY:
This was a single centre study comprised of two stages (Parts I and II). Part II was a 12 week randomised double blind comparison of Movicol and Lactulose Dry as maintenance therapy on an out-patient basis. The aim was to evaluate the safety and efficacy of Movicol in the treatment of faecal impaction in children

DETAILED DESCRIPTION:
Two days following disimpaction (Part I of the clinical trial) patients were assigned (based on their randomisation number) to receive either Movicol or Lactulose as maintenance therapy for the remainder of the study. At discharge all patients received the appropriate supply of study medication. This includes 1 week's overage should they miss their next visit to the ProMotion clinic. They did not know whether they have been randomised to receive Movicol or Lactulose Dry.

Following discharge patients were contacted after 3-5 days by telephone or home visit (whichever was appropriate) to encourage treatment and to ensure compliance. Parents were instructed to contact the Pro-Motion team who would advise appropriately if patients had any difficulty i.e. none, irregular and/ or uncomfortable or very loose bowel movements.

The daily use of Movicol or Lactulose Dry during Part II was recorded in the diary. If the dose of Movicol or Lactulose was changed by the Pro-Motion team at any time then it was documented appropriately in the patient notes and the case report form.

ELIGIBILITY:
Inclusion Criteria:

* patients that, in the opinion of the investigator, are constipated/faecally impacted as to require hospital stay to treat and/or relieve the impaction
* children aged 2 - 11 years old inclusive
* patients of either sex

Exclusion Criteria:

Patients with

* intestinal perforation or obstruction
* severe inflammatory conditions of the intestinal tract
* uncontrolled renal/hepatic/cardiac diseases
* uncontrolled endocrine disorder(s)
* any neuromuscular condition affecting bowel function
* hypersensitivity to lactulose or PEG or other constituent of Movicol
* patients who have taken any investigational drug in the three months
* patients or patients whose parents would in the opinion of the investigator are unable to comply with requirements of the study

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2000-10; Study Completion 2002-07

PRIMARY OUTCOMES:
compare the safety and efficacy of Movicol and Lactulose Dry as maintenance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David CA Candy, MD, Principal Investigator — St. Richard's Hospital
Locations (1):
- St Richard's Hospital, Royal West Sussex Hospital NHS Trust, Chichester, United Kingdom

REFERENCES:
- [Background] Dalziel SR et al. Efficacy of Movicol in children with faecal impaction. A series of en case histories (A13). British Society of Paediatric Gastroenterologists Annual Meeting. Bristol:21-22, Jan 2000
- [Background] Attar A, Lemann M, Ferguson A, Halphen M, Boutron MC, Flourie B, Alix E, Salmeron M, Guillemot F, Chaussade S, Menard AM, Moreau J, Naudin G, Barthet M. Comparison of a low dose polyethylene glycol electrolyte solution with lactulose for treatment of chronic constipation. Gut. 1999 Feb;44(2):226-30. doi: 10.1136/gut.44.2.226. PMID 9895382
- [Result] Candy DC, Edwards D, Geraint M. Treatment of faecal impaction with polyethelene glycol plus electrolytes (PGE + E) followed by a double-blind comparison of PEG + E versus lactulose as maintenance therapy. J Pediatr Gastroenterol Nutr. 2006 Jul;43(1):65-70. doi: 10.1097/01.mpg.0000228097.58960.e6. PMID 16819379